CLINICAL TRIAL: NCT05687877
Title: General Drug Use-Result Study of Evusheld Intramuscular Injection Set (Treatment and Prevention of Symptomatic Disease Caused by SARS-CoV-2 Infection)
Brief Title: Evusheld Japan PMS_Japan Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8850C00019
Record Dates: First submitted 2022-12-16; First posted 2023-01-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
To investigate intends to evaluate the incidence of adverse drug reactions (ADRs) in individuals who receive Evusheld in clinical practice to determine its post-marketing safety profile in Japanese.

DETAILED DESCRIPTION:
To investigate intends to evaluate the incidence of adverse drug reactions (ADRs) in individuals who receive Evusheld in clinical practice to determine its post-marketing safety profile in Japanese.

The investigation will be conducted as the addtional pharmacovigilance activitiy specified in the Japan Risk Management Plan (J-RMP) of Evusheld in compliance with the Ministerial Ordinance on Good Post-marketing Study Practice (GPSP Ordinance) and for the purpose of application for re-examination under Article 14-4 of the Act on Securing Quality, Efficacy and Safety of Products Including Pharmaceuticals and Medical Devices (PMD Act).

ELIGIBILITY:
Inclusion Criteria:

* For treatment of symptomatic disease caused by SARS-CoV-2 infection; Patients with risk factors for severe SARS-CoV-2 infection who do not require supplemental oxygen.
* For prevention of symptomatic disease caused by SARS-CoV-2 infection; Individuals for whom SARS-CoV-2 vaccination is not recommended OR those who are considered to have an inadequate response to a COVID-19 vaccine due to immunodeficiencies AND who is not close contacts such as family members or other people living in the same dwelling as patients infected with SARS-CoV-2.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment and prevention of symptomatic disease caused by SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs | 24weeks(6 months)
  The incidence of ADRs related to Evusheld Safety Specification; anaphylaxis and other serious allergic reactions, cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (18):
- Japan (18):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Nara
  - Research Site, Numakunai
  - Research Site, Osaka
  - Research Site, Tokyo
  - Research Site, Tottori

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.All request will be evaluated as per the AZ disclosure commitment.
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contact for data accessors ) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, Pleas review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00019&attachmentIdentifier=121b186c-aa89-4283-97e7-6b2ff27380bb&fileName=D8850C00019_Redacted_CSR_Synopsis.pdf&versionIdentifier=